CLINICAL TRIAL: NCT03991871
Title: HARapan kiTa ECP (External Counter Pulsation) Study HARTEC Study
Acronym: HARTEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Bambang Dwiputra, MD Cardiologist, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HARTEC Study
Record Dates: First submitted 2018-06-25; First posted 2019-06-19 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cardiac Rehabilitation; Angiogenesis; Refractory Angina
Keywords: Refractory Angina; Angiogenesis; External Counterpulsation; Angiopoietin
MeSH Terms: conditions — Angina Pectoris | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Comparison between two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): 35 hours ECP treatment, initial treatment pressure is 75 mmHg
  Interventions: Device: External Counter Pulsation (ECP) therapy
- Intervention Group (Experimental): 35 hours ECP treatment, initial treatment pressure is 300 mmHg
  Interventions: Device: External Counter Pulsation (ECP) therapy

INTERVENTIONS:
Device: External Counter Pulsation (ECP) therapy — 35 hours ECP treatment in 35 sessions

SUMMARY:
External Counterpulsation Therapy (ECP) is a therapeutic procedure that performed on patients with angina or heart failure to relieve the ischaemic symptoms, improve functional capacity, and quality of life. In recent studies, ECP has already proved to reduce angina symptoms, decrease degree of ischemic in heart train test. External Counterpulsation Therapy (ECP) therapy is a non-invasive technique for sequentially pressuring calf, lower thighs, and upper thighs through developed cuffs at pressure above systolic blood pressure when diastole, then deflated at systole.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of ECP therapy on cardiovascular hemodynamic, coronary perfusion, endothelial function, angiogenesis and artery genesis of the coronary blood vessel to refractory angina pectoris patients Refractory angina pectoris patients in Harapan Kita hospitals who do not respond to drugs adequately will be divided by 2 groups, control & treatment. Inclusion criteria include age 21 - 80 years, Refractory angina CCS III-IV whom are not candidate for Re-revascularization with proven data of: have stenosis on left main more than 50%, stenosis on main coronary right artery more than 70% or stenosis more than 70% on others vessels, conducted in coronary surgery conference with conservative decision (optimal medications).

Exclusion criteria include aorta aneurysm, abdominal aneurysm, acute coronary syndrome, acute heart failure, heavy aortic regurgitation, malignant arrhythmia, blood pressure above 180/100mmHg, acute limb ischemia, DVT, active thrombophlebitis, and pregnancy.

the investigator conducts a double-blind randomized control trial. The participants will get 35 hours ECP treatment, initial treatment pressure is 300 mmHg. whilst control groups will get 75mmHg. At the end of treatment, the investigator compare the hemodynamic effect on coronary perfusion, endothelial function, angiogenesis, and coronary blood vessel arteriogenesis. Quality of Life Improvement based on WHO-5 between groups

ELIGIBILITY:
Inclusion Criteria:

* age 21 - 80 years
* Refractory angina CCS III-IV whom are not candidate for Re-revascularization with proven data of: have stenosis on left main more than 50%, stenosis on main coronary right artery more than 70% or stenosis more than 70% on others vessels, conducted in coronary surgery conference with conservative decision (optimal medica mentosa).

Exclusion Criteria:

* aorta aneurysm,
* abdominalis aneurysm,
* acute coronary syndrome,
* acute heart failure,
* heavy aortic regurgitation,
* malignant arrhythmia,
* blood pressure above 180/100mmHg,
* acute limb ischaemia,
* DVT,
* active thrombophlebitis,
* pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Angiopoietin I concentration | 7 weeks
  hemodynamic effect on coronary perfusion. angiopoietin I involve in angiogenesis process. this study aims to investigate effects of External counterpulsation for refractory angina patients. it hypothesized to increase collateral artery which mechanism is by increasing angiogenesis process, measured with increase of Angiopoietin I and decrease of Angiopoietin II. Angiopoietin I level will be measured using ELISA technique.
MiRNA 92a concentration | 7 weeks
  microRNAs (miRNAs) are short (20-24 nt) non-coding RNAs that are involved in post-transcriptional regulation of gene expression in multicellular organisms by affecting both the stability and translation of mRNAs. miRNAs are transcribed by RNA polymerase II as part of capped and polyadenylated primary transcripts (pri-miRNAs) that can be either protein-coding or non-coding. The primary transcript is cleaved by the Drosha ribonuclease III enzyme to produce an approximately 70-nt stem-loop precursor miRNA (pre-miRNA), which is further cleaved by the cytoplasmic Dicer ribonuclease to generate the mature miRNA and antisense miRNA star (miRNA*) products. The mature miRNA is incorporated into a RNA-induced silencing complex (RISC), which recognizes target mRNAs through imperfect base pairing with the miRNA and most commonly results in translational inhibition or destabilization of the target mRNA. inhibition of MiRNA 92a prevents endothelial dysfunction.
Angiopoietin II concentration | 7 weeks
  Angiopoietin II established to play a role in blood vessel angiogenesis, antagonist of signaling through Tie2 tyrosine kinase receptor

SECONDARY OUTCOMES:
VEGFR-2 concentration | 7 weeks
  Vascular endothelial growth factor receptor-2 concentration, measured using ELISA
VEGF concentration | 7 weeks
  Vascular endothelial growth factor concentration, measured in plasma, using ELISA method
NT pro BNP concentration | 7 weeks
  Marker of heart failure. NTpro BNP will be measured pre and post external counterpulsation. BNP is actually produced primarily by the left ventricle of the heart (the heart's main pumping chamber). It is associated with blood volume and pressure and with the work that the heart must do in pumping blood throughout the body. Small amounts of a precursor protein, pro-BNP, are continuously produced by the heart. Pro-BNP is then cleaved by the enzyme called corin to release the active hormone BNP and an inactive fragment, NT-proBNP, into the blood.When the left ventricle of the heart is stretched, the concentrations of BNP and NT-proBNP produced can increase markedly. This situation indicates that the heart is working harder and having more trouble meeting the body's demands. This may occur with heart failure as well as with other diseases that affect the heart and circulatory system.
6 minute walking test distance (meters) | 7 weeks
  6 minutes walking test has long been known to measure functional capacity, will be measured pre and post ECP. 6-minutes walking test measuremet is in meter. it measure how far the participants could walk in 6 minutes.
NYHA Class index | 7 weeks
  New York Heart Association (NYHA) Functional Classification to classify severity of heart failure symptoms. It places patients in one of four categories based on how much they are limited during physical activity.
CCS Class index | 7 weeks
  Canadian Cardiovascular Society (CCS) classify angina symptoms into CCS class. it is to classify severity of angina symptoms. it places patients in one of four categories based on the severity of the angina on affecting and limiting phisical activity.
WHO 5 index | 7 weeks
  measuring quality of life, it will be measured pre and post ECP. The 5-item World Health Organization Well-Being Index (WHO-5) is among the most widely used questionnaires assessing subjective psychological well-being. Since its first publication in 1998, the WHO-5 has been translated into more than 30 languages and has been used in research studies all over the world. We now provide a systematic review of the literature on the WHO-5.

CONTACTS AND LOCATIONS:
Overall Officials: Ade Meidian Ambari, MD,FIHA, Principal Investigator — National Cardiovascular Center Harapan Kita Hospital Indonesia
Locations (1):
- Ade Meidian Ambari, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim MC, Kini A, Sharma SK. Refractory angina pectoris: mechanism and therapeutic options. J Am Coll Cardiol. 2002 Mar 20;39(6):923-34. doi: 10.1016/s0735-1097(02)01716-3. PMID 11897431
- [Result] Loh PH, Cleland JG, Louis AA, Kennard ED, Cook JF, Caplin JL, Barsness GW, Lawson WE, Soran OZ, Michaels AD. Enhanced external counterpulsation in the treatment of chronic refractory angina: a long-term follow-up outcome from the International Enhanced External Counterpulsation Patient Registry. Clin Cardiol. 2008 Apr;31(4):159-64. doi: 10.1002/clc.20117. PMID 18404725
- [Result] Henry TD, Satran D, Jolicoeur EM. Treatment of refractory angina in patients not suitable for revascularization. Nat Rev Cardiol. 2014 Feb;11(2):78-95. doi: 10.1038/nrcardio.2013.200. Epub 2013 Dec 24. PMID 24366073
- [Derived] Ambari AM, Lilihata G, Zuhri E, Ekawati E, Wijaya SA, Dwiputra B, Sukmawan R, Radi B, Haryana SM, Adiarto S, Hanafy DA, Zamroni D, Elen E, Mangkuanom AS, Santoso A. External Counterpulsation Improves Angiogenesis by Preserving Vascular Endothelial Growth Factor-A and Vascular Endothelial Growth Factor Receptor-2 but Not Regulating MicroRNA-92a Expression in Patients With Refractory Angina. Front Cardiovasc Med. 2021 Oct 25;8:761112. doi: 10.3389/fcvm.2021.761112. eCollection 2021. PMID 34760951